CLINICAL TRIAL: NCT01117376
Title: Methylnaltrexone vs Erythromycin for Facilitating Gastric Emptying Time in Critically Ill Patients Intolerant to Enteral Feeding
Brief Title: Methylnaltrexone vs Erythromycin for Facilitating Gastric Emptying Time in Critically Ill Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated because of unavailibility of Methylnaltrexone in the region
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: M. H. Dabbaghmanesh, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT-88-01-36-1601
Record Dates: First submitted 2010-04-30; First posted 2010-05-05 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2010-05

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Erythromycin; Methylnaltrexone; ICU
MeSH Terms: conditions — Gastroparesis | interventions — Erythromycin; methylnaltrexone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythromycin (Active Comparator): 21 patients admitted in ICU with intolerance to enteral feeding defined as more than 250 ml of gastric residual volume (GRV) found by aspiration technique.
  Interventions: Drug: Erythromycin
- Methylnaltrexone (Active Comparator): 21 patients admitted in ICU with intolerance to enteral feeding defined as more than 250 ml of gastric residual volume (GRV) found by aspiration technique.
  Interventions: Drug: Methylnaltrexone

INTERVENTIONS:
Drug: Erythromycin — Erythromycin 250 mg intravenous Q6h for 4 doses
  Arms: Erythromycin
Drug: Methylnaltrexone — Methylnaltrexone 12 mg subcutaneous Q12h for 2 doses
  Arms: Methylnaltrexone

SUMMARY:
42 patients admitted in ICU with intolerance to enteral feeding (GRV more than 250 ml) are recruited. All patients enter a primary acetaminophen absorption test study as baseline. Serum levels of acetaminophen will be measured by florescence polarization method at 15,30,45,60,90,120,180,240,480 minutes after enteral administration of 975 mg acetaminophen. Then the patients will be randomized to methylnaltrexone or erythromycin group.Another acetaminophen absorption test with the same schedule will be done after the last dose of each drug.The area under the curve for acetaminophen blood level will be used to compare the effect of two studied drugs on gastric emptying time.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in intensive care unit in a university affiliated hospital
* Receiving continuous enteral feeding through a nasogastric tube
* Gastric residual volume more than 250 ml checked by aspiration technique

Exclusion Criteria:

* Receiving the study drugs or metoclopramide within 24 hours of inclusion
* Known allergy to interventional drugs or acetaminophen
* Gastrointestinal bleeding or surgery on GI system within 24 hours of inclusion
* Crohn's disease
* GI perforation or obstruction
* Short bowel syndrome
* Liver failure or 2 of the followings:

  * Transaminase enzymes more than 3 times normal
  * Prothrombin time more than 2 times normal
  * Total bilirubin more than 3 times normal
* Patients on hemodialysis or CRRT
* Hemodynamically unstable patients including:

  * Mean arterial pressure less than 65 mmHg
  * Infusion of inotropes and vasopressors
  * Uncorrected acute blood loss; hemoglobin concentration less than 6.5 mg%.
* Documented or suspected pregnancy
* Obesity; actual body weight more than 1.5 times ideal body weight
* Myasthenia Gravis.
* Opioid drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying time | within 8 hours after drug administration
  to measure gastric emptying time within 8 hours after administration of either 4 doses of 250 mg intravenous erythromycin Q6h or 2 doses of methylnaltrexone 12 mg subcutaneous Q12h with acetaminophen absorption test method

SECONDARY OUTCOMES:
Tolerance to enteral feeding | 24 hours after intervention
  Tolerance to enteral feeding administered via nasogastric tube within 24 hours after administration of either erithromycin 250 mg intravenous Q6h or methylnaltrexone 12 mg subcutaneous Q12h.Gastric residual volume will be measured Q4h by aspiration method and if less than 250 ml would be considered as tolerance to enteral feeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemazee Hospital, Shiraz, Fars, Iran